CLINICAL TRIAL: NCT06265532
Title: Collagen-targeted PET Imaging for Assessment of EGCG Effect
Brief Title: Collagen-targeted Positron Emission Tomography (PET) Imaging for Assessment of EGCG Effect
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hal Chapman (Other)
Collaborators: Cornell University (Other); Massachusetts General Hospital (Other); University of Michigan (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Hal Chapman, Professor, Medicine, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00060157; R33HL158540 (NIH)
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — epigallocatechin gallate

STUDY DESIGN:
Intervention Model Description: This is an optional substudy to the phase I study: "Dose ranging study of oral epigallocatechin-3-gallate (EGCG) given daily for 12 weeks to patients with Idiopathic Pulmonary Fibrosis (IPF) evaluating safety, PK interactions with standard of care drugs, and biomarkers of drug effect." Up to twenty-two participants participating in the aforementioned study will be enrolled into this sub-study. This substudy will be conducted at a select number of sites with capabilities for performing [68Ga]CBP8 PET.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants will be on one of the standard of care drugs (nintedanib or pirfenidone) and blindly given EGCG or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- EGCG 300 mg (Active Comparator): Patients enrolled in this group will be given oral capsule EGCG 300 mg daily with doctor provided anti-fibrotic for 12 weeks.
  Interventions: Drug: EGCG 300 mg
- Placebo for EGCG 300 mg (Placebo Comparator): Patients enrolled in this group will be given oral capsule Placebo daily for 12 weeks with doctor provided anti-fibrotic. The number of placebo capsules will be equal to that of 300 mg EGCG.
  Interventions: Drug: Placebo for EGCG 300 mg
- EGCG 600 mg (Active Comparator): Patients enrolled in this group will be given oral capsule EGCG 600 mg daily with doctor provided anti-fibrotic for 12 weeks.
  Interventions: Drug: EGCG 600 mg
- Placebo for EGCG 600 mg (Placebo Comparator): Patients enrolled in this group will be given oral capsule Placebo daily for 12 weeks with doctor provided anti-fibrotic. The number of placebo capsules will be equal to that of 600 mg EGCG.
  Interventions: Drug: Placebo for EGCG 600 mg

INTERVENTIONS:
Drug: EGCG 300 mg — Participants will be administered EGCG as part of the phase I study: "Dose ranging study of oral epigallocatechin-3-gallate (EGCG) given daily for 12 weeks to patients with Idiopathic Pulmonary Fibrosis (IPF) evaluating safety, PK interactions with standard of care drugs, and biomarkers of drug effect."
  Other Names: Dietary Supplement: EGCG Capsules with EGCG (at least 94% purity). 300 mg EGCG (2 capsules) taken orally daily for 12 weeks.
  Arms: EGCG 300 mg
Drug: Placebo for EGCG 300 mg — Participants will be administered placebo for EGCG as part of the phase I study: "Dose ranging study of oral epigallocatechin-3-gallate (EGCG) given daily for 12 weeks to patients with Idiopathic Pulmonary Fibrosis (IPF) evaluating safety, PK interactions with standard of care drugs, and biomarkers of drug effect."
  Other Names: Dietary Supplement: Placebo Placebo (2 capsules) taken orally daily for 12 weeks.
  Arms: Placebo for EGCG 300 mg
Drug: EGCG 600 mg — Participants will be administered placebo for EGCG as part of the phase I study: "Dose ranging study of oral epigallocatechin-3-gallate (EGCG) given daily for 12 weeks to patients with Idiopathic Pulmonary Fibrosis (IPF) evaluating safety, PK interactions with standard of care drugs, and biomarkers of drug effect."
  Other Names: Dietary Supplement: EGCG Capsules with EGCG (at least 94% purity). 600 mg EGCG (4 capsules) taken orally daily for 12 weeks.
  Arms: EGCG 600 mg
Drug: Placebo for EGCG 600 mg — Participants will be administered placebo for EGCG as part of the phase I study: "Dose ranging study of oral epigallocatechin-3-gallate (EGCG) given daily for 12 weeks to patients with Idiopathic Pulmonary Fibrosis (IPF) evaluating safety, PK interactions with standard of care drugs, and biomarkers of drug effect."
  Other Names: Dietary Supplement: Placebo Placebo (4 capsules) taken orally daily for 12 weeks.
  Arms: Placebo for EGCG 600 mg

SUMMARY:
The primary purpose of this substudy is to determine if collagen-targeted PET using the type 1 collagen-targeted PET probe, Gallium-68 (68Ga)-labeled collagen binding probe 8 (CBP8) can inform as to drug effect of EGCG and assist in dose selection.

DETAILED DESCRIPTION:
This is an optional sub-study of the phase I study: "Dose ranging study of oral epigallocatechin-3-gallate (EGCG) given daily for 12 weeks to patients with Idiopathic Pulmonary Fibrosis (IPF) evaluating safety, pharmacokinetic (PK) interactions with standard of care drugs, and biomarkers of drug effect." Up to twenty-two participants participating in the aforementioned study will be enrolled into this sub-study. This substudy will be conducted at a select number of sites with capabilities for performing [68Ga]CBP8 PET.

Eligible participants who consent to the substudy will undergo [68Ga]CBP8 PET-CT or [68Ga]CBP8 PET-MRI at two time points. Participants will undergo 68Ga-CBP8 PET within 7 days prior to randomization and then again within 7 days prior to day 84 of the phase I study.

The hypothesis is that [68Ga]CBP8 PET will detect decreased collagen deposition in individuals treated with EGCG compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in and eligible (based on screening procedures - Visit 1) for the main EGCG Phase 1 study, "Dose ranging study of oral epigallocatechin-3-gallate (EGCG) given daily for 12 weeks to patients with Idiopathic Pulmonary Fibrosis (IPF) evaluating safety, PK interactions with standard of care drugs, and biomarkers of drug effect
2. Signed informed consent

Exclusion Criteria:

1. Pregnant or breastfeeding (a negative quantitative serum human chorionic gonadotropin (hCG) pregnancy test is required for females having child-bearing potential before the participant can participate)*
2. Research-related radiation exposure exceeds 50 millisievert (mSv) in the prior 12 months
3. Determined by the investigator to be clinically unsuitable for the study

Additional exclusion criteria for participants undergoing PET-MRI:

1. Electrical implants such as cardiac pacemaker, defibrillator, or perfusion pump
2. Metallic or electric implants contraindicated for magnetic resonance-PET (MR-PET) scanning
3. Claustrophobic reactions
4. Estimated glomerular filtration rate (eGFR) of less than 30 mL/min/1.73 m2 within the prior 30 days
5. Known allergy to gadolinium

   * Women of childbearing potential (WCBP) are defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 24 consecutive months if < 55 years or 12 months if ≥ 55 years.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Change in collagen probe uptake over the entire lungs | From baseline to 12 weeks
  Changes in lung collagen uptake will be measured using the PET probe [68]Ga-CBP8. Measurements will be made over the entire lungs using standardized uptake values.

OTHER OUTCOMES:
Change in peak enhancement over the entire lungs | From baseline to 12 weeks
  Changes in peak enhancement will be measured using dynamic-contrast enhanced MRI. This exploratory outcome is only relevant for participants that undergo PET/MRI.
Change in the rate of contrast washin over the entire lungs | From baseline to 12 weeks
  Changes in rate of contrast washin will be measured using dynamic-contrast enhanced MRI. This exploratory outcome is only relevant for participants that undergo PET/MRI.
Change in the area under the curve at 60 seconds over the entire lungs | From baseline to 12 weeks
  Changes in the area under the curve at 60 seconds will be measured using dynamic-contrast enhanced MRI. This exploratory outcome is only relevant for participants that undergo PET/MRI.
Change in the full width at half maximum over the entire lungs | From baseline to 12 weeks
  Changes in the full width at half maximum will be measured using dynamic-contrast enhanced MRI. This exploratory outcome is only relevant for participants that undergo PET/MRI.
Change in the rate of contrast washout over the entire lungs | From baseline to 12 weeks
  Changes in the rate of contrast washout will be measured using dynamic-contrast enhanced MRI. This exploratory outcome is only relevant for participants that undergo PET/MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Martinez, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Montesi SB, Izquierdo-Garcia D, Desogere P, Abston E, Liang LL, Digumarthy S, Seethamraju R, Lanuti M, Caravan P, Catana C. Type I Collagen-targeted Positron Emission Tomography Imaging in Idiopathic Pulmonary Fibrosis: First-in-Human Studies. Am J Respir Crit Care Med. 2019 Jul 15;200(2):258-261. doi: 10.1164/rccm.201903-0503LE. No abstract available. PMID 31161770
- [Result] Izquierdo-Garcia D, Desogere P, Fur ML, Shuvaev S, Zhou IY, Ramsay I, Lanuti M, Catalano OA, Catana C, Caravan P, Montesi SB. Biodistribution, Dosimetry, and Pharmacokinetics of 68Ga-CBP8: A Type I Collagen-Targeted PET Probe. J Nucl Med. 2023 May;64(5):775-781. doi: 10.2967/jnumed.122.264530. Epub 2022 Dec 8. PMID 37116909